CLINICAL TRIAL: NCT04967703
Title: Effect of Radial Shock Wave and Ultrasound Therapy Combined With Traditional Physical Therapy Exercises on Foot Function and Dorsiflexion Range in Plantar Fasciitis: A Prospective Randomized Clinical Trial
Brief Title: Physiotherapy Protocols in Treating Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Jouf University (Other)
Responsible Party: Principal Investigator, Khaled Z. Fouda, Associate Professor of Physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-13-S-071(068)
Record Dates: First submitted 2021-07-07; First posted 2021-07-19 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Plantar Fascitis
Keywords: plantar fasciitis; foot function index; ultrasound; radial shock wave
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasound therapy protocol (Experimental): Patients in group A received ultrasound therapy protocol with the following parameters (1 MHz frequency, intensity of 1.5 W/cm2 and use of continuous mode of ultrasound for 5 minutes).
  Interventions: Procedure: Group A
- Radial shock wave therapy protocol (Experimental): Patients in group B received radial shock wave therapy protocol with the following parameters: (1) the energy level was 0.12 mJ/mm2 equivalent to 2.5 bar intensity, (2) the number of shoots was 2000, (3) the frequency was 8 Hz.
  Interventions: Procedure: Group B
- Combined therapy protocol (Experimental): Patients in group C received a combination of both ultrasound therapy and radial shock wave therapy protocol.
  Interventions: Procedure: Group C

INTERVENTIONS:
Procedure: Group A — Patients received ultrasound therapy protocol with the following parameters (1 MHz frequency, intensity of 1.5 W/cm2 and use of continuous mode of ultrasound for 5 minutes), in addition to a conventional physiotherapy program consisting of calf muscles stretching, plantar fascia stretch, strengthening exercises and manual massage for 3 sessions per week, for 4 weeks
  Other Names: Ultrasound therapy protocol
  Arms: Ultrasound therapy protocol
Procedure: Group B — Patients received radial shock wave therapy protocol with the following parameters (1) the energy level was 0.12 mJ/mm2 equivalent to 2.5 bar intensity, (2) the number of shoots was 2000, (3) the frequency was 8 Hz, in addition to the same conventional physiotherapy program given for group A
  Other Names: Radial shock wave therapy protocol
  Arms: Radial shock wave therapy protocol
Procedure: Group C — Patients received both ultrasound and radial shock wave therapy, in addition to the same conventional physiotherapy program given for group A
  Other Names: Combined therapy protocol
  Arms: Combined therapy protocol

SUMMARY:
This study aimed to investigate the efficacy of different physical therapy protocols in the treatment of chronic plantar fasciitis patients. Patients in this study were randomly assigned into 3 groups. Group A received ultrasound therapy protocol, group B received radial shock wave therapy protocol and group C received a combination of both ultrasound therapy and radial shock wave therapy protocol. All patients were also received a traditional physical therapy program. Foot function was evaluated by foot function index and ankle dorsiflexion range of motion was measured by Baseline® bubble inclinometer at the baseline and 4 weeks after treatment

DETAILED DESCRIPTION:
Sixty nine patients having unilateral chronic plantar fasciitis will be recruited for the study from Al-Qurayyat General Hospital, in Al-Jouf Region, Saudi Arabia. The inclusion criteria were as follows: patients suffered planter fasciitis of more than 3 months, maximum tenderness near the medial calcaneal insertion and pain was greater than 4 on visual analogue scale during taking the first steps in the morning. Patients were excluded if they had previous ankle or foot surgery or pathology, or if they had a previous history of shock wave therapy or topical corticosteroid injections to the ankle or foot, circulatory disturbances in the lower extremities, neuropathic or radicular pain in the lower limbs. Participants with systemic diseases that cause foot discomfort, such as ankylosing spondylitis, psoriatic arthritis, rheumatoid arthritis, and gout, as well as those with type I or type II diabetes and pregnancy, were also excluded from the study.

The patients were randomly assigned into 3 equal groups (n = 23). Group A received ultrasound therapy protocol using Enraf Nonius Sonoplus 490, Netherlands. Group B received radial shock wave therapy protocol using Swiss DolorClast® Master, Electro Medical Systems, SA, Nyon, Switzerland. Group C received a combination of both ultrasound therapy and radial shock wave therapy protocol. All patients also received a traditional physical therapy program (3 sessions per week, for 4 weeks) consisting of Calf muscles stretching and plantar fascia stretching. Foot function and Ankle dorsiflexion range of motion were evaluated at the baseline and 4 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffered plantar fasciitis of more than 3 months
* Maximum tenderness near the medial calcaneal insertion and pain was greater than 4 on visual analogue scale during taking the first steps in the morning

Exclusion Criteria:

* Bilateral plantar fasciitis
* Previous ankle or foot surgery or pathology
* If they had a previous history of shock wave therapy or topical corticosteroid injections to the ankle or foot
* Circulatory disturbances in the lower extremities
* Neuropathic or radicular pain in the lower limb
* Participants with systemic diseases that cause foot discomfort, such as ankylosing spondylitis, psoriatic arthritis, rheumatoid arthritis, and gout, as well as those with type I or type II diabetes and pregnancy, were also excluded from the study.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Foot function | From baseline to 4 weeks after treatment
  A modified version of the original foot function index was used to assess the change in foot function

SECONDARY OUTCOMES:
Ankle dorsiflexion range of motion | From baseline to 4 weeks after treatment
  A Baseline® bubble inclinometer was used to assess the change in Ankle dorsiflexion range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Z. Fouda, PhD, Principal Investigator — Associate Professor of Physical Therapy
Locations (1):
- Al Qurayyat General Hospital, Qurayyat, Jouf Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared including a summary of the results after the study completion date.
Supporting Information: Study Protocol
Time Frame: The dead time for IPD will be 30 June. 2024
Access Criteria: will be uploaded on the official site of CTR
URL: https://www.europeanreview.org/article/32287

REFERENCES:
- See also: Free Full Paper — https://www.europeanreview.org/article/32287
- Available data/document: Full Paper — http://www.europeanreview.org/article/32287